CLINICAL TRIAL: NCT00499031
Title: A Phase II Evaluation of Cetuximab (Erbitux®, C225, NSC# 714692) in the Treatment of Persistent or Recurrent Squamous or Non-Squamous Cell Carcinoma of the Cervix
Brief Title: Cetuximab in Treating Patients With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0227E; NCI-2009-00596 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BMS-CA225-275; CDR0000554455; GOG-0227E (Other: Gynecologic Oncology Group); GOG-0227E (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Cervical Squamous Cell Carcinoma; Recurrent Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cetuximab

ARMS (1):
- Treatment (cetuximab) (Experimental): Patients receive cetuximab IV over 120 minutes on day 1.
  Interventions: Biological: Cetuximab

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Chimeric MoAb C225; Erbitux; IMC-C225

SUMMARY:
This phase II trial is studying cetuximab to see how well it works in treating patients with persistent or recurrent cervical cancer. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of cetuximab for patients with persistent or recurrent carcinoma of the cervix.

II. To determine the frequency of patients who survive progression-free for at least 6 months after initiating therapy or have objective tumor response.

SECONDARY OBJECTIVES:

I. To characterize the distribution of progression-free survival and overall survival.

II. To determine the effect of cetuximab on the duration of objective response in persistent or recurrent carcinoma of the cervix.

III. To determine the nature and degree of toxicity of cetuximab as assessed by CTCAE v3.0 in this cohort of patients.

OUTLINE:

Patients receive cetuximab IV over 120 minutes on day 1. Courses repeat once weekly in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed (with physical exams and histories) every three months for the first two years and then every six months for the next three years.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Patients must have persistent or recurrent squamous or non-squamous cell carcinoma of the cervix with documented disease progression (disease not amenable to curative therapy)

    * Histologic documentation of the original primary tumor is required via the pathology report
  * All patients must have measurable disease defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded)

    * Each lesion must be ≥ 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT scan, and MRI, OR ≥ 10 mm when measured by spiral CT scan
  * Patients must have at least one target lesion to be used to assess response on this protocol

    * Tumors within a previously irradiated field will be designated as nontarget lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
  * Patients must have had one prior systemic chemotherapeutic regimen for management of advanced, metastatic, or recurrent carcinoma of the cervix

    * Chemotherapy administered in conjunction with primary radiation as a radiosensitizer is not counted as a systemic chemotherapy regimen
  * Patients must not be eligible for a higher priority GOG protocol, if one exists

    * In general, this would refer to any active GOG phase III protocol for the same patient population
* Exclusion criteria:

  * Patients with craniospinal metastases
* Inclusion criteria:

  * Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2 or patients who have received two prior regimens must have a GOG performance status of 0 or 1
  * Patients should be free of active infection requiring antibiotics
  * Platelet count ≥ 100,000/μl
  * ANC ≥ 1,500/μl
  * Creatinine ≤ 1.5 x institutional upper limit normal (ULN)
  * Bilirubin ≤ 1.5 x ULN
  * SGOT and alkaline phosphatase ≤ 2.5 x ULN
  * Neuropathy (sensory and motor) ≤ CTCAE v3.0 grade 1
  * Calcium < 11.0 mg/dL
  * Patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiating protocol therapy and be practicing an effective form of contraception during protocol therapy and for at least two months following completion of protocol therapy
* Exclusion criteria:

  * Patients with a history of other invasive malignancies, with the exception of nonmelanoma skin cancer and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last five years

    * Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
  * Patients who have a significant history of cardiac disease (i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure, or uncontrolled arrhythmias) within 6 months of registration
  * Patients who have an uncontrolled seizure disorder or active neurological disease
  * Patients known to be seropositive for HIV and active hepatitis, even if liver function studies are in the eligible range
  * Pregnant or nursing women or women of childbearing potential unless using effective contraception as determined by the investigator
  * Known hemorrhagic diathesis or active bleeding disorder
* Inclusion criteria:

  * Recovery from effects of recent surgery, radiotherapy, or chemotherapy

    * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration (continuation of hormone replacement therapy is permitted)
    * Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration
  * Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent cervical disease according to the following definition:

    * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
  * Patients must not have received any non-cytotoxic therapy for management of recurrent or persistent cervical disease
  * Patients must not be receiving any other investigational agent
* Exclusion criteria:

  * Patients who have received prior therapy with cetuximab or any other anti-epidermal growth factor receptor antibody
  * Patients who have received any prior therapy with a tyrosine kinase inhibitor that targets the EGFR pathway
  * Patients who have received prior chimerized or murine monoclonal antibody therapy
  * Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis other than for the treatment of cervical cancer within the last five years are excluded

    * Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration and the patient remains free of recurrent or metastatic disease
  * Patients who have received prior chemotherapy for any abdominal or pelvic tumor other than for the treatment of cervical cancer within the last five years are excluded

    * Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration and that the patient remains free of recurrent or metastatic disease
  * Patients who have undergone major surgery, excluding diagnostic biopsy, within 30 days (to allow for full recovery) prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-06; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Santin, Principal Investigator — Gynecologic Oncology Group
Locations (22):
- United States (22):
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Decatur Memorial Hospital, Decatur, Illinois
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Singing River Hospital, Pascagoula, Mississippi
  - CoxHealth South Hospital, Springfield, Missouri
  - Island Gynecologic Oncology, Brightwaters, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cetuximab): Day 1: 400 mg/m2 loading dose of cetuximab IV over 120 minutes; Day 8 and weekly thereafter: 250 mg/m2 cetuximab IV over 60 minutes (one cycle = four weeks) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Treatment (Cetuximab)
Started | 38 (Total number participants enrolled on study)
Completed | 35 (Total number participants that are eligible and evaluable.)
Not Completed | 3
Not completed — Improper pre-protocol treatment | 1
Not completed — Required test not done | 1
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: Total number eligible and evaluable participants
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 35
Age, Customized [Mean (Standard Deviation); unit: years] | 49.7 (9.3)
Age, Customized [Number; unit: participants]
  30-39 years | 3
  40-49 years | 16
  50-59 years | 10
  60-69 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
Cell Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 4
  Mixed Epithelial Carcinoma | 1
  Adenosquamous | 6
  Squamous Cell Carcinoma | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Greater Than 6 Months
Time Frame: At 6 months
Population: Total number of eligible and evaluable participants
Measure: Number; unit: participants
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 35
participants
  No | 30
  Yes | 5

2. Primary Outcome: Objective Tumor Response Assessed by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Response is measured according to Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.0):
  Complete Response (CR) is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart.
  Partial Response (PR) is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  Disease Progression is at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
  Stable Disease is any condition not meeting the above criteria.
  Indeterminate is defined as having no repeat tumor assessments following initiation of study therapy for reasons unrelated to symptoms or signs of disease.
Time Frame: every other cycle for the first 6 months; then every 3 months x 2; then every 6 months
Population: Total number of eligible and evaluable participants
Measure: Number; unit: participants
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 35
participants
  Stable disease | 11
  Disease progression | 23
  Indeterminate | 1

3. Secondary Outcome: Duration of Progression-free Survival
Time Frame: From study entry until disease progression, death or date of last contact, up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Objective Response Rate
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Frequency and Severity of Adverse Effects as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Duration of Overall Survival
Time Frame: From study entry to death or the date of last contact, up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study entry until disease progression or study withdrawal. Patients will then be monitored for delayed toxicity for a 5 year period.
Description: From protocol activation through Sept. 30, 2010, Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (CTCAE v3.0) are utilized for defining and grading specific adverse events reported through the AdEERS system. As of Oct. 1, 2010, CTCAE v 4.0 will be utilized for AE reporting. AEs are reported in ClinicalTrials.gov using CTCAE v3.0.
Arm/Group | Treatment (Cetuximab)
Serious Adverse Events (participants affected / at risk) | 15/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cetuximab) (N=35)
Inr (Vascular disorders) | 1
Fever (General disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 3
Fistula, Gi - Rectum (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain - Other (General disorders) | 1
Pain: Back (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cetuximab) (N=35)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1
Rhinitis (Immune system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 4
Platelets (Blood and lymphatic system disorders) | 5
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 10
Lymphopenia (Blood and lymphatic system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 26
Weight Gain (General disorders) | 1
Fever (General disorders) | 2
Weight Loss (General disorders) | 5
Fatigue (General disorders) | 20
Death No Ctcae Term - Death Nos (General disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 2
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 23
Dry Skin (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3
Flushing (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 2
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 1
Incontinence, Anal (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 2
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Stomach (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 15
Anorexia (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 7
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 1
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 2
Hemorrhage, Gi - Stomach (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Esophagus (Infections and infestations) | 1
Febrile Neutropenia (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lip/Perioral (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Conjunctiva (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 1
Inf Unknown Anc: Oral Cavity-Gums (Infections and infestations) | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 1
Edema: Limb (Blood and lymphatic system disorders) | 4
Ast (Metabolism and nutrition disorders) | 3
Creatinine (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Ggt (Metabolism and nutrition disorders) | 2
Alt (Metabolism and nutrition disorders) | 2
Alkaline Phosphatase (Metabolism and nutrition disorders) | 5
Bilirubin (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 10
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 12
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 3
Mood Alteration - Anxiety (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 3
Neuropathy-Motor (Nervous system disorders) | 1
Watery Eye (Eye disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 1
Blurred Vision (Eye disorders) | 2
Pain - Other (General disorders) | 2
Pain: Urethra (General disorders) | 1
Pain: Pelvis (General disorders) | 2
Pain: Vagina (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 2
Pain: Throat/Pharynx/Larynx (General disorders) | 2
Pain: Head/Headache (General disorders) | 5
Pain: Neck (General disorders) | 1
Pain: Extremity-Limb (General disorders) | 5
Pain: Back (General disorders) | 7
Pain: Joint (General disorders) | 2
Pain: Bone (General disorders) | 1
Pain: Kidney (General disorders) | 1
Pain: Pain Nos (General disorders) | 1
Pain: Stomach (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 9
Pain: Face (General disorders) | 1
Pain: Muscle (General disorders) | 1
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Urinary Color Change (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 3
Vaginal Discharge (Reproductive system and breast disorders) | 2
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No